CLINICAL TRIAL: NCT02820675
Title: Quality Improvement in Infection COntrol and Sepsis Management in MOdel Regions / Deutsches Qualitaetsbuendnis Sepsis (German Quality Network Sepsis)
Brief Title: Quality Improvement in Infection COntrol and Sepsis Management in MOdel Regions
Acronym: icosmos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Sepsis Control and Care, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Vivantes Berlin Hospitals (Unknown); Klinikum Nürnberg (Other); Sana Clinics (Unknown); University Hospital Augsburg (Other); Zentralklinik Bad Berka (Other); Bundeswehrkrankenhaus Berlin (Other); University Hospital, Bonn (Other); Bremen Hospitals (Unknown); Herzzentrum Coswig (Other); Klinikum Lippe Detmold (Other); Krankenhaus Dresden Friedrichstadt (Unknown); Krankenhaus Düren (Unknown); Heinrich-Heine University, Duesseldorf (Other); Klinikum St. Georg gGmbH (Other); Rudolf Elle Hospital Eisenberg (Unknown); Klinikum Emden (Other); BG Klinikum Frankfurt Main (Unknown); SRH Hospital Gera (Unknown); Asklepios Clinics (Unknown); Greifswald University Hospital (Unknown); Deutsches Rotes Kreuz DRK-Blutspendedienst Baden-Wurttemberg-Hessen (Other); University Hospital in Halle (Other); Hannover Medical School (Other); University Hospital Schleswig-Holstein (Other); St. Elisabeth Hospital Cologne (Unknown); Leipzig University Hospital (Unknown); Magdeburg University Hospital (Unknown); Mannheim University Hospital (Unknown); Munich University Hospital Rechts der Isar (Unknown); Trauma Center Murnau (Unknown); Havelland Hospitals (Unknown); Nordhausen South Harz Hospital (Unknown); Oldenburg Hospital (Unknown); Rostock Southern City Hospital (Unknown); Saarbruecken Hospital (Unknown); Siegen Diakonie Hospital (Unknown); Stuttgart Hospital (Unknown); SRH Central Hospital Suhl (Unknown); MediClin Mueritz Hospital Waren (Unknown); Werdau Pleissetal Hospital (Unknown)
Responsible Party: Principal Investigator, Hendrik Rüddel, trial manager, leader of trial management team, Center for Sepsis Control and Care, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CSCCGermany
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: quality improvement; routine data; risk adjustment; sepsis, severe sepsis, septic shock; quality of coding
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention (Other): all hospitals participating in the icosmos trial will be supported in implenatation of the two main interventions.
  Interventions: Other: structured case analysis; Other: strucured screening "every patient, every shift"

INTERVENTIONS:
Other: structured case analysis — implementation of a structured analysis of cases coded as sepsis, severe sepsis, or septic shock after risk adjustment for low-risk-fatalities, high-risk-survivors, and coding errors for preventable deaths, best practice, quality improvement and improvement in coding precision.
Other: strucured screening "every patient, every shift" — implementation of a strutured screening and rescue algorithm on regular wards, emergency departements, and intermediate and intensive care units by checking every patient in every shifts for clinical signs of deterioration and apllying a rescue algorithm including consiliary help and/or the help of outreach teams

SUMMARY:
The German Quality Network Sepsis is an association trying to improve quality of care for patients with sepsis, severe sepsis and septic shock or being in risc thereof.

The icosmos trial investigates the impact on the use of routine data, a risk adjustment algorithm and feedback to all hospitals as well as a structured implementation for regular screening for deteriorating patients, and education on in-hospital mortality.

DETAILED DESCRIPTION:
All German hospitals provide a set of routine data to federal adminsitration for reimbursement. This dataset includes all ICD-10-Codes (German adaption) as well as all procedure codes.

This dataset is pseudonomized and risk adjusted for every individual case and afterwards feedbacked to each participating hospital including all accumulated data from all other hospitals as well as the German Average for sepsis mortalities provided by the German Federal Institute of Statistcs for benchmarkings.

Based on this data, the icosmos trial will provide support to all participating hospitals for two major strategies to be implemented

1. An algorithm for structured analysis of

   1. low-risk-fatalities as potentially preventable deaths for underlying problems in diagnosis, treatment, etc
   2. high-risk-survivors as "best practice"
   3. coding errors for improvement of coding quality
2. a structured sreening program of every patient on every ward in every shift for deterioration and support algorithms including consiliary support and outreach teams as well as structured education

The icosmos trial will investigate the effects as well on quality of coding and sepsis incidence as well as on sepsis-related sepsis in-hospital mortality for participating hospitals in comparison to the German Average.

ELIGIBILITY:
Inclusion Criteria for hospitals:

* hospitals willing to participate

Inclusion Criteria for patients / patients' data

* age over 16
* coding of sepsis, severe sepsis, septic shock

Exclusion Criteria for hospitals:

* no intensive care unit on site

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | 3 years
  in-hospital mortality of all patients coded with sepsis, severe sepsis and septic shock in absolute numbers and in relation to the German average
sepsis codings | 3 years
  developement of coding of sepsis, severe sepsis and septic shock in absolte numbers and in relation to the German Average

CONTACTS AND LOCATIONS:
Locations (1):
- CSCCGermany, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Our trial uses publicly accessible routine data and a risk adjustment algorithm being prepared for publication

REFERENCES:
- [Derived] Schwarzkopf D, Ruddel H, Grundling M, Putensen C, Reinhart K. The German Quality Network Sepsis: study protocol for the evaluation of a quality collaborative on decreasing sepsis-related mortality in a quasi-experimental difference-in-differences design. Implement Sci. 2018 Jan 18;13(1):15. doi: 10.1186/s13012-017-0706-5. PMID 29347952
- See also: trial homepage (in German) — http://www.icosmos.uniklinikum-jena.de